CLINICAL TRIAL: NCT01813682
Title: Effect of Iron-fortified TPN on Preterm Infants Anemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: qingya tang (Other)
Responsible Party: Sponsor-Investigator, qingya tang, profecer, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: eoitopia
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Preterm Infants
Keywords: preterm infant; anemia; iron fortified TPN
MeSH Terms: conditions — Premature Birth; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (No Intervention): preterm infants of this group with iron-free TPN for more than ten days, compare serum iron, iron protein, total iron binding force, MDA, 8-iso-PGF2α on baseline and after intervention.
- treatment group1 (Experimental): preterm infants of this group with iron supplementation of 200μg/kg/d for more than ten days, compare serum iron, iron protein, total iron binding force, MDA, 8-iso-PGF2α on baseline and after intervention.
  Interventions: Other: treatment group1
- treatment group2 (Experimental): preterm infants of this group with iron supplementation of 400μg/kg/d for more than ten days, compare serum iron, iron protein, total iron binding force, MDA, 8-iso-PGF2α on baseline and after intervention.
  Interventions: Other: treatment group2

INTERVENTIONS:
Other: treatment group1 — fe-1 group with TPN of iron supplementation of 200μg/kg/d.
  Arms: treatment group1
Other: treatment group2 — fe-2 group with TPN of iron supplementation of 400μg/BW (BW=birth weight)
  Arms: treatment group2

SUMMARY:
The purpose of this study is to determine whether iron-fortified TPN is effective in the preventative and treatment of preterm infants. Preterm infants are at risk for anemia especially in preterm infants. Generally the smaller Birth weight and gestational age the higher anemia rate in infants. About 25% to 85% of preterm infants develop evidence of anemia during infancy，77% VLBW（very low birth weight） infants developed anemia during the hospital stay. The effects of iron deficiency are pervasive and involve multiple organ systems. Poor physical growth, gastrointestinal disturbances, thyroid dysfunction, altered immunity and temperature instability has been attributed to iron deficiency in very low birth weight infants. So it is important to provide iron for preterm infants.

As enteral nutrition is not feasible soon after birth in most preterm infants, Parenteral iron administration is an efficacious method for us to select. For most preterm infants the use of TPN(total parenteral nutrition) is very common during the first ten days of life, so we hypothesis that iron-fortified TPN may have a preventative and treatment effect on preterm infants using TPN as a supplementation of oral nutrition; Iron-fortified TPN(total parenteral nutrition) can also improve iron store status of preterm infants. The higher concentration of iron used in this study the larger preventative or treatment effect on preterm infants anemia; It is safe to add Small dose of iron agent to TPN.

DETAILED DESCRIPTION:
Preterm infants are at high risk of anemia especially low birth weight infants, so it is important to supply iron with infants of this group.

90 preterm infants BW(birth weight) less than 2kg,entered neonatal intensive care unit(NICU) less than 72 hours and meet the Inclusion Criteria of this study will be Randomly divided into three groups, control group、 treatment group1 (200μg/kg/d,and the highest concentration of iron is ≤0.8g/100ml TPN)、treatment group2 （400μg/kg/d,and the highest concentration of iron is ≤0.8g/100ml TPN）. iron supplementation period for more than ten days. For three groups, complete blood counts, differential counts, and reticulocyte counts were measured weekly in samples obtained, serum iron, iron protein, total iron binding force were measured at baseline and after 2 weeks. Through comparative analysis of three groups, to find iron-fortified TPN whether affect anemia rate and iron storage in preterm. we also selected malondialdehyde (MDA)and 8-iso-prostaglandin F2α(8-iso-PGF2α) as our concerns about iron used in TPN induces oxidative stress index.

Iron protein determination use radioimmunoassay method, serum iron and total iron binding force determination use chemical method, MDA and 8-iso-PGF2α determination use enzyme-linked immunosorbent assay method.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with birth weight less than 2kg Have parenteral nutrition indication With written informed consent of parents or guardian

Exclusion Criteria:

* have already used TPN before randomization Kidney and liver function abnormal have hemolytic disease have hemorrhagic disease have Serious congenital malformation have septicemia have plethora newborn use TPN less than ten days

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
anemia rate | up to 2 weaks
  compare the anemia rate of three groups and identify the effect of iron-fortified TPN for preterm infants.

SECONDARY OUTCOMES:
iron status | baseline and more than ten days
  Serum iron, iron protein and total iron binding force are parameters used to test the effectiveness of iron-fortified TPN used for preterm infants.

OTHER OUTCOMES:
Oxidative stress parameters Oxidative stress parameters Oxidative stress parameters | baseline and more than ten days
  we use MDA、 8-iso-prostaglandin F2α as the oxidative stress parameters to identify the safety of iron-fortified TPN used in preterm infants.

CONTACTS AND LOCATIONS:
Overall Officials: qingya tang, M.D., Principal Investigator — Shanghai jiaotong university affiliated xinhua hospital
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China